CLINICAL TRIAL: NCT03855644
Title: Establishment for Prediction Model of Intraoperative Blood Transfusion for Patients With Pelvic Fracture in China: A Multicenter Observational Study
Brief Title: Blood Transfusion Among Patients With Pelvic Fracture in China
Acronym: PBM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other); Zhejiang Provincial People's Hospital (Other); Central South University (Other); Qilu Hospital of Shandong University (Other); Beijing Aerospace General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SXKThirdXiangyaHCSU
Record Dates: First submitted 2019-01-25; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Pelvic Fracture; Transfusion Reaction; Blood Transfusion Complication
Keywords: Pelvic Fracture; Predictive Model; Blood Transfusion; Perioperative period
MeSH Terms: conditions — Hip Fractures; Transfusion Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic fracture patients: (1) 1<Age<80, and Chinese residents living in China more than 3 years; (2) Hemoglobin value less than 100g/L during hospitalization; Not suffered from pelvic fracture within 3 months; Not suffer from pathological fractures of the pelvis caused by malignant tumors; without chronic anemia and coagulopathy; accept blood transfusion

SUMMARY:
According to the patient's blood management concept, this study intends to collect basic information, surgical data, blood transfusion related data and patient prognosis data of patients with pelvic fractures, and to construct a predictive model of intraoperative blood transfusion in patients with pelvic fractures by multiple linear regression analysis. To guide physicians use blood accurately during surgery. Prompt doctors to reduce blood transfusion dose and improve patient prognosis by stopping bleeding and blood recovery before surgery.

DETAILED DESCRIPTION:
2.1 Research Objectives: This study aims to construct a blood transfusion model for pelvic fractures, to guide the rational use of blood during surgery, and to improve the prognosis of patients.

2.2 Research content: 2.2.1 Collect basic data, surgical data, blood transfusion related data and patient prognosis related data of patients with pelvic fractures.

2.2.2 Gradually incorporate and exclude data from multiple linear regression models.

2.2.3 Verify the specificity and sensitivity of the intraoperative blood transfusion prediction model.

2.2.4 Create a visualization window to guide clinical blood. 2.2.5 Put into clinical trial and feedback, and continue to verify 2.3 Key issues to be resolved 2.3.1 The factors related to intraoperative blood transfusion in patients with pelvic fractures (such as blood oxygenation, blood loss, HB value, intraoperative autologous blood recovery, blood pressure, heart rate, etc.) were initially screened by univariate analysis.

2.3.2 Reasonably standardize the objective and subjective indicators of different units and different institutions.

2.4 Expected research results Intraoperative blood transfusion prediction model and window for patients with pelvic fractures.

2.5 Assessment indicators Published 1-2 papers. Create a visual applet and put it into trial.

ELIGIBILITY:
Inclusion Criteria:

* (1) 1<Age<80, and Chinese residents living in China more than 3 years;
* (2) Hemoglobin value less than 100g/L during hospitalization;

Exclusion Criteria:

* (1) Participants who suffered from pelvic fracture within 3 months
* (2) Participants who suffer from pathological fractures of the pelvis caused by malignant tumors
* (3) Participants with chronic anemia and coagulopathy
* (4) Participants who rufuse blood transfusion

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pelvic fractures who meet the standard in China, 1<Age<80.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-04-05 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Matta Radiographic Scoring | 6 months of postoperation
  Reductions were graded by the maximal displacement measured on the 3 standard views of the pelvis. Criteria were: excellent 4 mm or less, good 5 to 10 mm, fair 10 to 20 mm, and poor more than 20 mm.
Mortality | 24 hours after the Patients' Hospitalization
  Mortality during hospitalization

SECONDARY OUTCOMES:
Hb difference | 24 hours after transfusion
  Hb difference before and after transfusion
Pain assessed by the VAS | 15 minutes, 30 minutes, 1 hours, 2 hours, 4 hours, 6 hours, 12 hours, 18 hours, 24 hours postoperatively
  Change in the Pain Intensity Score (0-10 NRS)
Postoperative Duration of Stay in Hospital of patients | 52 Weeks
  The postoperative duration of stay in hospital of patients between the restrictive transfusion group and the liberal transfusion group are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sathy AK, Starr AJ, Smith WR, Elliott A, Agudelo J, Reinert CM, Minei JP. The effect of pelvic fracture on mortality after trauma: an analysis of 63,000 trauma patients. J Bone Joint Surg Am. 2009 Dec;91(12):2803-10. doi: 10.2106/JBJS.H.00598. PMID 19952241
- [Background] Perkins ZB, Maytham GD, Koers L, Bates P, Brohi K, Tai NR. Impact on outcome of a targeted performance improvement programme in haemodynamically unstable patients with a pelvic fracture. Bone Joint J. 2014 Aug;96-B(8):1090-7. doi: 10.1302/0301-620X.96B8.33383. PMID 25086126
- [Background] Santana-Cabrera L, Rodriguez Gonzalez F, Palacios MS. Delayed perforation of the sigmoid colon following a major pelvic fracture. J Emerg Trauma Shock. 2010 Oct;3(4):425-6. doi: 10.4103/0974-2700.70770. No abstract available. PMID 21063578
- [Background] Carson JL, Terrin ML, Noveck H, Sanders DW, Chaitman BR, Rhoads GG, Nemo G, Dragert K, Beaupre L, Hildebrand K, Macaulay W, Lewis C, Cook DR, Dobbin G, Zakriya KJ, Apple FS, Horney RA, Magaziner J; FOCUS Investigators. Liberal or restrictive transfusion in high-risk patients after hip surgery. N Engl J Med. 2011 Dec 29;365(26):2453-62. doi: 10.1056/NEJMoa1012452. Epub 2011 Dec 14. PMID 22168590
- [Background] Nathens AB. Massive transfusion as a risk factor for acute lung injury: association or causation? Crit Care Med. 2006 May;34(5 Suppl):S144-50. doi: 10.1097/01.CCM.0000214309.95032.65. PMID 16617259
- [Background] Ohmori T, Matsumoto T, Kitamura T, Tamura R, Tada K, Inoue T, Hayashi T, Numoto K, Tokioka T. Scoring system to predict hemorrhage in pelvic ring fracture. Orthop Traumatol Surg Res. 2016 Dec;102(8):1023-1028. doi: 10.1016/j.otsr.2016.09.007. Epub 2016 Nov 17. PMID 27865687
- [Background] Hardy JF, de Moerloose P, Samama CM; Members of the Groupe d'Interet en Hemostase Perioperatoire. Massive transfusion and coagulopathy: pathophysiology and implications for clinical management. Can J Anaesth. 2006 Jun;53(6 Suppl):S40-58. doi: 10.1007/BF03022251. PMID 16766790